CLINICAL TRIAL: NCT02137902
Title: Healing and Empowering Alaskan Lives Towards Healthy-Hearts Study
Acronym: HEALTHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); Alaska Native Tribal Health Consortium (Other); University of Alaska Anchorage (Other); Norton Sound Health Corporation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Judith Prochaska, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29638; 1R01HL117736 (NIH)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Tobacco Dependence
Keywords: Tobacco dependence; Cardiovascular disease; Risk behaviors; Smoking; Physical activity; Alaska Native people
MeSH Terms: conditions — Tobacco Use Disorder; Cardiovascular Diseases; Risk-Taking; Smoking; Motor Activity | interventions — Tobacco Products; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobacco/Physical Activity Intervention (Experimental): Includes a psychosocial component that utilizes a counselor-facing computer-assisted intervention with tailored counseling feedback focused on increasing intrinsic motivation, goal setting for tobacco and physical activity, adherence with nicotine replacement therapy, and self-monitoring with a pedometer-based walking program. The intervention will provide 12 weeks of nicotine replacement therapy for participants.
  Interventions: Behavioral: Tobacco/Physical Activity Intervention
- Diet plus BP/CHOL Intervention (Experimental): Consists of a psychosocial component that includes counselor-facing computer-assisted intervention with tailored counseling feedback focused on increasing intrinsic motivation, goal setting for managing hypertension and hypercholesterolemia, and adherence with antihypertensives and statins with supportive dietary changes. The intervention provides a cookbook of heart healthy regional recipes and medication bag for storing medications.
  Interventions: Behavioral: Diet plus BP/CHOL Intervention

INTERVENTIONS:
Behavioral: Tobacco/Physical Activity Intervention — Telemedicine stage-tailored counseling intervention focused on increasing intrinsic motivation and goal setting for tobacco and physical activity, adherence with nicotine replacement therapy (NRT, patch plus gum or lozenge), and self-monitoring with a pedometer-based walking program.
  Arms: Tobacco/Physical Activity Intervention
Behavioral: Diet plus BP/CHOL Intervention — Telemedicine stage-tailored counseling intervention focused on increasing intrinsic motivation, goal setting for managing HTN and HCL, and adherence with antihypertensives and statins with supportive dietary changes. Includes a native diet cookbook and medication bag.
  Arms: Diet plus BP/CHOL Intervention

SUMMARY:
This study aims to identify effective and cost-effective interventions for tobacco use and other risk behaviors for cardiovascular disease among Alaska Native people in rural villages. In a randomized controlled trial, the study will compare interventions using telemedicine to promote the American Heart Association's identified ideal health behaviors (nonsmoking and physical activity) relative to ideal health factors (managing cholesterol and blood pressure).

DETAILED DESCRIPTION:
In an RCT, we will compare 2 active treatments delivered over 12-months via telehealth services linking participants in rural villages to Anchorage and Stanford-based study counselors overcoming access-to-care for CV preventive health issues. The village AN health aides will facilitate data collection and telehealth connectivity. Intervention contacts occur at baseline, 3-, 6- and 12-months follow-up, with the final assessment at 18-months. The repeated intervention contacts provide iterative computerized feedback reflecting prior responses and encouragement of adoption and maintenance of behavioral health goals. The groups are:

1. Tobacco/Physical Activity Intervention (n=150), consisting of a psychosocial component that includes counselor-facing computer-assisted intervention with tailored counseling feedback focused on increasing intrinsic motivation, goal setting for tobacco and physical activity, adherence with nicotine replacement therapy (NRT, patch plus gum or lozenge), and self-monitoring with a pedometer-based walking program. The study will provide 12-weeks of NRT for participants randomized to this intervention condition.
2. HTN/HCL (HTN/HC, n=150), consisting of a psychosocial component that includes counselor-facing computer-assisted intervention with tailored counseling feedback focused on increasing intrinsic motivation, goal setting for managing HTN and HCL, and adherence with antihypertensives and statins with supportive dietary changes. The AN health plan covers antihypertensive and statins as a benefit to patients and would be prescribed as part of standard of care (i.e., not prescribed for the purposes of this research); however, strategies to maximize medication adherence are needed, hence the focus of this intervention.

The counseling and print materials are highly individualized, unique to the participant, thereby minimizing the likelihood of cross-condition contamination, determined to be minimal in prior investigations. For the research study, participant eligibility criteria include AN heritage; daily cigarette smoking; and hypertension, hyperlipidemia, or established vascular disease. Intention to change the targeted risk behaviors will not be required to participate. Utilizing telemedicine technology and Transtheoretical Model-tailored interventions, the trial aims to reach at-risk AN people regardless of residential location or current motivation. The primary outcome is biochemically-confirmed tobacco abstinence using anabasine. Secondary outcomes include moderate-to-vigorous physical activity assessed by self-report, blood pressure, cholesterol ratio, medication adherence, dietary change, body mass index, Framingham index, multibehavioral impact factor, a linear index, and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Smoking > 5 cigarettes/day and > 100 cigarettes in one's lifetime
* Hypertension, hypercholesterolemia, or established vascular disease
* Fluent in English language

Exclusion Criteria:

* Dementia or other brain injury
* Pregnancy or breastfeeding
* Currently engaged in tobacco treatment or using cessation pharmacotherapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2015-06-01; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Smoking Status: 7-day point prevalence abstinence | Assessed at baseline, 3, 6, 12, and 18 months
  Change from baseline as no tobacco use, including a puff, in the past 7 days

SECONDARY OUTCOMES:
Minutes of moderate-to-vigorous physical activity in past 7 days | Assessed at baseline, 3, 6, 12, and 18 months
  self-reported minutes of moderate-to-vigorous physical activity
Blood pressure | Assessed at baseline, 3, 6, 12, and 18 months
  Measured as systolic/diastolic in mmHg
Total, LDL, and HDL cholesterol | Assessed at baseline and 18 months
  measured in milligrams per deciliter of blood (mg/dL)
Body Mass Index (BMI) | Assessed at baseline, 3, 6, 12, and 18 months
  weight (in kilograms) over height squared (in centimeters)
Framingham Risk Factor Score | Assessed at baseline and 18 months
  gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual
Medication Adherence | Assessed at baseline, 3, 6, 12 and 18 months
  self-reported assessment of adherence to BP and CHOL meds
Dietary Quality | Assessed at baseline, 3, 6, 12 and 18 months
  culturally tailored FFQ assessing consumption of native and non-native foods
Multiple Risk Behavior Change Impact Factor | Assessed at baseline, 3, 6, 12 and 18 months
  intervention efficacy times participation summed over the multiple behavioral targets, I = ∑# of behaviors(n) (En × Pn)
Linear index of multiple behavior change | Assessed at baseline, 3, 6, 12 and 18 months
  computed by subtracting baseline scores from follow-up scores for each risk behavior, dividing by the standard deviation of the difference (i.e., z-score), and summing across the individual risks (smoking, exercise, diet, adherence)

CONTACTS AND LOCATIONS:
Overall Officials: Judith J Prochaska, PhD, MPH, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Norton Sound Health Corporation, Nome, Alaska
  - Stanford Hospital and Clinics, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prochaska JJ, Benowitz NL. The Past, Present, and Future of Nicotine Addiction Therapy. Annu Rev Med. 2016;67:467-86. doi: 10.1146/annurev-med-111314-033712. Epub 2015 Aug 26. PMID 26332005
- [Background] Prochaska JJ, Benowitz NL. Smoking cessation and the cardiovascular patient. Curr Opin Cardiol. 2015 Sep;30(5):506-11. doi: 10.1097/HCO.0000000000000204. PMID 26196657
- [Derived] Prochaska JJ, Epperson A, Skan J, Oppezzo M, Barnett P, Delucchi K, Schnellbaecher M, Benowitz NL. The Healing and Empowering Alaskan Lives Toward Healthy-Hearts (HEALTHH) Project: Study protocol for a randomized controlled trial of an intervention for tobacco use and other cardiovascular risk behaviors for Alaska Native People. Contemp Clin Trials. 2018 Aug;71:40-46. doi: 10.1016/j.cct.2018.06.003. Epub 2018 Jun 2. PMID 29864548

DOCUMENTS (1):
  • Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT02137902/ICF_000.pdf